CLINICAL TRIAL: NCT07071571
Title: Evaluation of the Usability and Safety of the Newly Developed Piezoelectric Sensor Intraoperative Nerve Monitoring Device in Thyroid and Parathyroid Surgery: A Pilot Study
Brief Title: New Intraoperative Nerve Monitoring Device
Acronym: IONM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Erhan Aysan, Prof Dr, SB Istanbul Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 111.023; No any fund (Other: No any fund)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Thryoid Cancer; parathyrıoid Adenoma
Keywords: neuromonitorization; introperative; recurrent nerve; new device

STUDY DESIGN:
Intervention Model Description: Recurrent nerve monitoring will be performed in patients with thyroid or parathyroid surgery indications.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thyro,d cases (Active Comparator)
  Interventions: Device: neuromonitoring

INTERVENTIONS:
Device: neuromonitoring — new neuromonitorin device will use

SUMMARY:
This study is testing a new device developed to protect the recurrent laryngeal nerve, which is at risk of damage during thyroid and parathyroid surgeries.

DETAILED DESCRIPTION:
This study is testing a new device developed to protect the recurrent laryngeal nerve, which is at risk of damage during thyroid and parathyroid surgeries. Such devices are still used in surgical routine, but research has been initiated on this subject due to the higher sensitivity and reliability of this new device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70, diagnosis of benign/malignant thyroid disease, informed consent

Exclusion Criteria:

* History of previous nerve injury, concomitant neurological disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
recurrent nerve identification | introperatively
  nerve will be identified with new device

IPD SHARING:
Plan to Share IPD: No
No need